CLINICAL TRIAL: NCT00443014
Title: Phase 4 Study of Cognitive Therapy and Donepezil in Alzheimers Disease.
Brief Title: The Dementia Study in Northern Norway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: County Officer of Nordland, Moloveien 2, 8006 Bodø, Norway (Unknown); Norwegian Foundation for Health and Rehabilitation (Other); Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 200201054-12/12BMA2/400
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Alzheimer Disease
Keywords: Stimulation therapy; Acetylcholinesterase inhibitors; Synergetic
MeSH Terms: conditions — Alzheimer Disease | interventions — Physical Examination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Cognitive stimulation therapy (Experimental): Patients with recently diagnosed dementia in five of the study municipality.
  Interventions: Device: Cognitive, physical and social stimulation
- B Care as usual (No Intervention)

INTERVENTIONS:
Device: Cognitive, physical and social stimulation — Sessions of 30 minutes daily five days a week for one year
  Arms: A Cognitive stimulation therapy

SUMMARY:
The Dementia Study in Northern Norway is an open controled intervention trial carried out in nine rural municipalities, five of which allocated to intervention and four to control. A RCT with donepezil and placebo is superimposed on all patients included in the study. In this way the study has a 2x2 factorial design. The outcome measures are changes in cognitive performance and ADL function measured by standardized cognitive and neuropsychological tests every four months during a one-year follow-up.

The main goal of this study is to examine the effect of systematically and individually adjusted stimulation therapy on cognitive function in patients having recent diagnoses of Alzheimer´s disease (AD).

A secondary goal is to examine whether or not ChEI has an additional effect on cognitive function superimposed on stimulation therapy.

From January 2006 to 31th March 2008 187 patients with a recent diagnosis of dementia were included. Patients were recruited by GPs in routine practice (n=87) and by a population based screening (n=100).Screening recruited younger patients with a higher MMSE-score, and relatively more men. All over, women were older and at a more serious disease stage. After age adjusting significantly more women were living single and required more supports from the community nursery.

DETAILED DESCRIPTION:
Nine municipalities with 11807 inhabitants 65 years and older were allocated to intervention or control, five and four municipalities in each group, respectively. A panel of psychiatric nurses, university lecturers and members of the competence centre of dementia in Northern Norway have worked out a program of stimulation therapy adjusted to each participant taking the stage of functional impairment, education level and work experience into consideration. The individual stimulation program is selected and implemented, based on the life history for each patient, and carried out for a minimum of 30 minutes 5 days a week in the intervention group, as compared to the control group receiving routine care. The individual stimulation program was monitored and adjusted during the period of intervention. All patients included in the nine municipalities were randomized to donepezil or placebo in a double blind manner.

Consequently, the present study has a double design; - an open prospective non-pharmaceutical intervention with control group, to which a double blind and randomized placebo-controlled trial is superimposed (2x2 factorial design). Each patient have been followed-up for one year. The clinical period was three years, two of them allocated recruitment and the third to secure a one-year intervention for all participants.

The Progress of the Study The recruitment of patients through routine general practice has not been successful. The participating general practitioners (GP) rarely examined patients suffering from cognitive impairment. Sometimes patients with a presumptive diagnosis of dementia were prescribed cholinesterase inhibitors (ChEI) without a preceding clinical examination. As a result of this lack of corporation only 27 patients were recruited to the study during the first year. During the subsequent six months some of the nine participating municipalities reorganized their caring routines for patients suffering from dementia. More patients were examined and diagnosed and another 60 patients were recruited to the study.

As a consequence of the unsatisfactory progress in recruiting patients to the study by GPs in routine clinical practice, the study protocol was changed and the recruiting procedures were supplemented by a population-based screening. The study population (65 years+) was invited to attend the survey by responding to and return a postal questionnaire containing five simple questions regarding memory and cognitive deficits. The screening program was accomplished in June 2007 with a response rate of approximately 32 % for self-reported memory deficits. An algorithm categorizes the responders. Those belonging to the category with the highest risk of having a diagnosis of dementia were invited to a clinical examination carried out by physicians from the study administration. Those fulfilling the inclusion criteria were then asked to be included in this Dementia Study in Northern-Norway.

More than 700 responders answered NO to the five questions about cognitive impairment but YES to a question about participating in the study. From this group of presumptively cognitive healthy people we randomly draw a sample of 500 persons who was invited to participate in a control group for the AD participants. Of these 200 individuals were confirmed cognitively healthy and included in the control group. The two groups have been compared according to clinical data, co-morbidity and drug consumption. A biobank containing whole blood, plasma and serum from AD participants and the cognitively healthy control group is established.

The stimulation program was executed as presupposed, and the randomisation procedures and administration of the medical treatment (placebo/donepezil) has been accomplished without any problems.

The following papers have been published in BMC Methodology and in BMC Geriatrics:

http://www.biomedcentral.com/1471-2318/11/58

http://www.biomedcentral.com/1471-2288/10/35

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 65-94 years with a recent diagnosed AD and without any contraindications for the use of donepezil.
* A MMSE sum score has to be at least10 points

Exclusion Criteria:

* Behavioural disturbance which make cooperation and cognitive testing impossible.
* Individuals with reduced approval competence expressing any reluctance to participate are excluded, as well as those not understanding the purpose of the study and who have relatives or care givers disapproving participation.
* Individuals having a diagnosis of dementia treated with CheI at entry are also excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 187 (Actual)
Dates: Start 2003-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The cognitive function is measured with the Alzheimer's Disease Assessment | Every fourth month in one year

SECONDARY OUTCOMES:
Changes in Activity of Daily Living (ADL) measured by standardized tests. | When the patient is included and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Fred Andersen, MD GP, Principal Investigator — University of Northern Norway; Torgeir Engstad, MD, PhD, Study Director — University of Northern Norway
Locations (1):
- Arran Lulesami Centre, Drag, Nordland, Norway

REFERENCES:
- [Background] Graff MJ, Vernooij-Dassen MJ, Thijssen M, Dekker J, Hoefnagels WH, Rikkert MG. Community based occupational therapy for patients with dementia and their care givers: randomised controlled trial. BMJ. 2006 Dec 9;333(7580):1196. doi: 10.1136/bmj.39001.688843.BE. Epub 2006 Nov 17. PMID 17114212
- [Derived] Andersen F, Viitanen M, Halvorsen DS, Straume B, Wilsgaard T, Engstad TA. The effect of stimulation therapy and donepezil on cognitive function in Alzheimer's disease. A community based RCT with a two-by-two factorial design. BMC Neurol. 2012 Jul 19;12:59. doi: 10.1186/1471-2377-12-59. PMID 22813231
- [Derived] Andersen F, Engstad TA, Straume B, Viitanen M, Halvorsen DS, Hykkerud S, Sjobrend K. Recruitment methods in Alzheimer's disease research: general practice versus population based screening by mail. BMC Med Res Methodol. 2010 Apr 29;10:35. doi: 10.1186/1471-2288-10-35. PMID 20429946
- See also: Related Info — http://dsnn.no